CLINICAL TRIAL: NCT04147117
Title: Cervical Pessary to Prevent Preterm Singleton Birth in High Risk Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC-35-17
Record Dates: First submitted 2019-10-16; First posted 2019-10-31 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Preterm Birth
Keywords: Preterm Birth; Cervical Pessary; Obstetrical history; Cervical length
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pessary Group (Experimental): A pessary certified is inserted through the vagina with the woman in recumbent position and is placed around the cervix.
  Correct placement of the pessary is assessed by ultrasound. Patients on the pessary group are specially awarded about adverse symptoms and the need of immediate report in case of pain, bleeding and symptomatic contractions.
  The pessary is not removed when symptoms of infection occur after pessary insertion, but appropriate treatment is given.
  The pessary is removed at 37 weeks of pregnancy. Indications for pessary removal before 37 weeks are: active vaginal bleeding, premature labor not responding to tocolysis or severe patient discomfort.
  Interventions: Device: Cervical pessary
- Control group (No Intervention): Current management for the follow-up of these women in the PBPC.

INTERVENTIONS:
Device: Cervical pessary — Cervical pessary is a silicone ring with a smaller diameter to be fitted around the cervix and a larger diameter to fix the device to the pelvic floor. It modifies the direction of the cervix to the posterior vaginal wall.
  Arms: Pessary Group

SUMMARY:
DESIGN: Observational prospective study. INCLUSION CRITERIA: All women are 18 years old of age or older with high risk for preterm birth, based on clinical history, and between 18.0 weeks and 23.6 weeks of pregnancy. SAMPLE SIZE: 214 asymptomatic high risk pregnant women.

METHODOLOGY: Patient selection, obtaining of informed consent, randomization for cervical placement of pessary. Current follow-up until delivery. Pessary is removed at 37 week or before in some specific situations.

MAIN OUTCOME: sPTB <370 weeks of gestation. SECONDARY OUTCOMES: Pregnancy outcomes and a neonatal composite morbidity. EXPECTED RESULTS: Cervical pessary reduces sPB below 37 weeks in high risk of preterm birth population.

DETAILED DESCRIPTION:
Spontaneous preterm birth (sPB) is still a leading cause of neonatal and infant death and responsible of neonatal morbidity as cerebral palsy. In spite of improvements of neonatal care, rates of preterm birth have not changed in the recent 10 years.

Clinical risk factors for preterm birth include: 1) Demographic characteristics such a low socioeconomic status, poor antenatal care, malnutrition or extremes in maternal age; 2) Behavioral factors including smoking, illicit drug abuse, alcohol consumption or heavy physical work; 3) Obstetric history including uterine malformation, previous preterm labor or preterm rupture of membranes (PROM), previous cervical surgery, late miscarriage >16-17 weeks; 4) Aspects of the current pregnancy as multiple pregnancy, genital tract bleeding or infection, Preterm Rupture of Membranes (PROM), short cervix and others.

In nulliparous women with no previous pregnancies or fetal losses >16 weeks, screening based on clinical history (maternal racial origin, age, height, smoking status and method of conception) could detect about 20% of sPB. In women with previous pregnancies at or beyond 16 weeks the detection rate is doubled by incorporating obstetric history.

The risks for women with a previous spontaneous preterm birth with a normal cervix in pregnancy are not negligible. It has been suggested that there is a continuum risk dependent on absolute cervical length while other authors showed that absolute length of cervix above 25mm had little impact on the risk of preterm birth before 35 weeks. A posterior study has not identified any clinical or obstetric risk factors in high-risk women with cervical length greater than 25mm that could help to identify those who will subsequently have a spontaneous preterm birth.

The risk of preterm birth is inversely related to cervical length (CL) as measured by ultrasound. Current options for the management of short cervix in singleton pregnancies are: vaginal progesterone, with proved benefit; cervical cerclage in high risk and short cervix, and cervical pessary.

Cervical pessary is a silicone ring with a smaller diameter to be fitted around the cervix and a larger diameter to fix the device to the pelvic floor. It modifies the direction of the cervix to the posterior vaginal wall.

Three randomized trials involving women with singleton low risk pregnancies and short cervix provided controversial results regarding the effect of cervical pessary on the rate of sPB before 34 weeks; in one trial, involving 380 women, the rate of this outcome was significantly lower with a pessary than with no pessary (6% vs 27%); in another trial, involving 108 women, there was no significant effect (9.4% vs 5.5%, respectively) and in the largest trial, involving 935 women, no benefits were found (12.9% vs 11.3%, respectively).

Nowadays high-risk population with normal cervix is managed by cervical length surveillance and physical activity restriction, as progesterone has not a proved benefit in women at risk because of previous history but normal cervix.

Cervical pessary has not been tested specifically in high risk population. In PECEP study a total number of 42 patients (11% of each group) had at least one previous preterm birth. Authors did not report differences in the risk of preterm birth before 34 weeks in this subgroup. In Nicolaides study, 154 patients had previous birth before 37 weeks: 70 were treated with pessary and 84 with expectant management. The reported risk of birth before 34 weeks was 10.1% and 19.5%, respectively. In spite of the increased risk in expectant group, these differences were not significant (OR 0.47 (0.18-1.21) p= 0.12). In both trials, women included has short cervix.

Even that group of women with previous preterm birth were included in the previous trials, pessary has not been proved in a specific group of population with previous history of preterm birth or uterine-cervical factors. Therefore, there is a lack of information in this topic.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Age > 18 years old.
* Gestational age between 18.0 -23.6 weeks of gestation.
* Asymptomatic singleton pregnancies, with at least one of the following:

  * Previous spontaneous preterm delivery or PPROM (23 - 34.6 weeks).
  * Previous spontaneous second trimester miscarriage (16.0-22.6 weeks).
  * Previous surgery on uterine cervix.
  * Uterine malformation.
* Able to sign informed consent form.

Exclusion Criteria:

* Congenital, chromosomal abnormalities or stillbirth in current pregnancy before randomization.
* Women with an obstetrical history of iatrogenic preterm birth indicated for maternal or fetal conditions.
* Symptomatic high-risk women or preterm prelabor rupture of membranes (PROM) in the current pregnancy.
* Pregnant women with an indication of prophylactic cervical cerclage due to her own obstetrical history.
* Pregnant women with an indication to perform a cervical cerclage, prior to study inclusion.
* Cerclage in situ.
* Active vaginal bleeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Spontaneous preterm birth before 37 weeks of gestation | 3 years
  Delivery < 37.0 weeks of gestation (Yes/No)

SECONDARY OUTCOMES:
Preterm birth 34 weeks | 5 months
  Birth before 34 weeks of gestation (Yes/No)
Preterm birth 28 weeks | 5 months
  Birth before 28 weeks of gestation (Yes/No)
PPROM before 34 weeks | 5 months
  Preterm premature rupture of membranes before 34 weeks (Yes/No)
Threatened preterm labor | 5 months
  Number of admissions for threatened preterm labor <34weeks of gestation
Cervical trauma | 5 months
  Serious cervical or vaginal trauma (Yes/No)
Pessary tolerance | 5 months
  Intolerance to pessary (Yes/No)
Infection | 5 months
  Vaginal infection (Yes/No)
Progesterone co-treatment | 5 months
  Need for progesterone co-treatment (Yes/No)
Choriomanionitis | 5 months
  Clinical chorioamnionitis (Yes/No)
Maternal mortality or morbidity | 5 months
  Maternal mortality or severe morbidity (Yes/No)
Neonatal birthweight | 5 months
  Birth weight in grams
Neonatal outcomes APGAR | 5 months
  5 min APGAR score < 7 (Yes/No)
Neonatal outcomes umbilical artery pH | 5 months
  Umbilical artery pH at delivery <7.1 (Yes/No)
Neonatal outcomes NICU | 5 months
  Need for NICU admission (Yes/No)
Neonatal outcomes for respiratory support | 5 months
  Need for respiratory support (Yes/No)
Neonatal outcomes SDR | 5 months
  Respiratory distress syndrome (Yes/No)
Neonatal outcomes IVH | 5 months
  Intraventricular haemorrhage (Yes/No)
Neonatal outcomes NEC | 5 months
  Necrotizing enterocolitis (Yes/No)
Neonatal outcomes. Death | 5 months
  Neonatal death (Yes/No)
Neonatal outcomes. Sepsis | 5 months
  Neonatal sepsis (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Irene Ferrero Martínez, MD,PhD, Principal Investigator — BCNatal | Hospital Sant Joan de Déu - Hospital Clínic; Montse Palacio Riera, MD,PhD, Study Director — BCNatal | Hospital Clínic- Hospital Sant Joan de Déu
Locations (1):
- Hospital Sant Joan de Déu. BCNatal | Barcelona Center for Maternal Fetal and Neonatal Medicine | Hospital Clínic - Hospital Sant Joan de Déu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beta J, Akolekar R, Ventura W, Syngelaki A, Nicolaides KH. Prediction of spontaneous preterm delivery from maternal factors, obstetric history and placental perfusion and function at 11-13 weeks. Prenat Diagn. 2011 Jan;31(1):75-83. doi: 10.1002/pd.2662. PMID 21210482
- [Background] Sotiriadis A, Papatheodorou S, Kavvadias A, Makrydimas G. Transvaginal cervical length measurement for prediction of preterm birth in women with threatened preterm labor: a meta-analysis. Ultrasound Obstet Gynecol. 2010 Jan;35(1):54-64. doi: 10.1002/uog.7457. PMID 20014326
- [Background] Celik E, To M, Gajewska K, Smith GC, Nicolaides KH; Fetal Medicine Foundation Second Trimester Screening Group. Cervical length and obstetric history predict spontaneous preterm birth: development and validation of a model to provide individualized risk assessment. Ultrasound Obstet Gynecol. 2008 May;31(5):549-54. doi: 10.1002/uog.5333. PMID 18432605
- [Background] Owen J, Szychowski JM, Hankins G, Iams JD, Sheffield JS, Perez-Delboy A, Berghella V, Wing DA, Guzman ER; Vaginal Ultrasound Trial Consortium. Does midtrimester cervical length >/=25 mm predict preterm birth in high-risk women? Am J Obstet Gynecol. 2010 Oct;203(4):393.e1-5. doi: 10.1016/j.ajog.2010.06.025. Epub 2010 Aug 12. PMID 20708169
- [Background] Care AG, Sharp AN, Lane S, Roberts D, Watkins L, Alfirevic Z. Predicting preterm birth in women with previous preterm birth and cervical length >/= 25 mm. Ultrasound Obstet Gynecol. 2014 Jun;43(6):681-6. doi: 10.1002/uog.13241. PMID 24186101
- [Background] Romero R, Nicolaides K, Conde-Agudelo A, Tabor A, O'Brien JM, Cetingoz E, Da Fonseca E, Creasy GW, Klein K, Rode L, Soma-Pillay P, Fusey S, Cam C, Alfirevic Z, Hassan SS. Vaginal progesterone in women with an asymptomatic sonographic short cervix in the midtrimester decreases preterm delivery and neonatal morbidity: a systematic review and metaanalysis of individual patient data. Am J Obstet Gynecol. 2012 Feb;206(2):124.e1-19. doi: 10.1016/j.ajog.2011.12.003. Epub 2011 Dec 11. PMID 22284156
- [Background] Berghella V, Mackeen AD. Cervical length screening with ultrasound-indicated cerclage compared with history-indicated cerclage for prevention of preterm birth: a meta-analysis. Obstet Gynecol. 2011 Jul;118(1):148-155. doi: 10.1097/AOG.0b013e31821fd5b0. PMID 21691173
- [Background] Owen J, Hankins G, Iams JD, Berghella V, Sheffield JS, Perez-Delboy A, Egerman RS, Wing DA, Tomlinson M, Silver R, Ramin SM, Guzman ER, Gordon M, How HY, Knudtson EJ, Szychowski JM, Cliver S, Hauth JC. Multicenter randomized trial of cerclage for preterm birth prevention in high-risk women with shortened midtrimester cervical length. Am J Obstet Gynecol. 2009 Oct;201(4):375.e1-8. doi: 10.1016/j.ajog.2009.08.015. PMID 19788970
- [Background] Abdel-Aleem H, Shaaban OM, Abdel-Aleem MA. Cervical pessary for preventing preterm birth. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD007873. doi: 10.1002/14651858.CD007873.pub3. PMID 23728668
- [Background] Goya M, Pratcorona L, Merced C, Rodo C, Valle L, Romero A, Juan M, Rodriguez A, Munoz B, Santacruz B, Bello-Munoz JC, Llurba E, Higueras T, Cabero L, Carreras E; Pesario Cervical para Evitar Prematuridad (PECEP) Trial Group. Cervical pessary in pregnant women with a short cervix (PECEP): an open-label randomised controlled trial. Lancet. 2012 May 12;379(9828):1800-6. doi: 10.1016/S0140-6736(12)60030-0. Epub 2012 Apr 3. PMID 22475493
- [Background] Hui SY, Chor CM, Lau TK, Lao TT, Leung TY. Cerclage pessary for preventing preterm birth in women with a singleton pregnancy and a short cervix at 20 to 24 weeks: a randomized controlled trial. Am J Perinatol. 2013 Apr;30(4):283-8. doi: 10.1055/s-0032-1322550. Epub 2012 Aug 8. PMID 22875662
- [Background] Nicolaides KH, Syngelaki A, Poon LC, de Paco Matallana C, Plasencia W, Molina FS, Picciarelli G, Tul N, Celik E, Lau TK, Conturso R. Cervical pessary placement for prevention of preterm birth in unselected twin pregnancies: a randomized controlled trial. Am J Obstet Gynecol. 2016 Jan;214(1):3.e1-9. doi: 10.1016/j.ajog.2015.08.051. Epub 2015 Aug 28. PMID 26321037
- [Background] Orzechowski KM, Boelig RC, Berghella V. Cervical Length Screening in Asymptomatic Women at High Risk and Low Risk for Spontaneous Preterm Birth. Clin Obstet Gynecol. 2016 Jun;59(2):241-51. doi: 10.1097/GRF.0000000000000195. PMID 27015227
- [Background] O'Brien JM, Adair CD, Lewis DF, Hall DR, Defranco EA, Fusey S, Soma-Pillay P, Porter K, How H, Schackis R, Eller D, Trivedi Y, Vanburen G, Khandelwal M, Trofatter K, Vidyadhari D, Vijayaraghavan J, Weeks J, Dattel B, Newton E, Chazotte C, Valenzuela G, Calda P, Bsharat M, Creasy GW. Progesterone vaginal gel for the reduction of recurrent preterm birth: primary results from a randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2007 Oct;30(5):687-96. doi: 10.1002/uog.5158. PMID 17899572
- [Background] DeFranco EA, O'Brien JM, Adair CD, Lewis DF, Hall DR, Fusey S, Soma-Pillay P, Porter K, How H, Schakis R, Eller D, Trivedi Y, Vanburen G, Khandelwal M, Trofatter K, Vidyadhari D, Vijayaraghavan J, Weeks J, Dattel B, Newton E, Chazotte C, Valenzuela G, Calda P, Bsharat M, Creasy GW. Vaginal progesterone is associated with a decrease in risk for early preterm birth and improved neonatal outcome in women with a short cervix: a secondary analysis from a randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2007 Oct;30(5):697-705. doi: 10.1002/uog.5159. PMID 17899571
- [Background] Dodd JM, Jones L, Flenady V, Cincotta R, Crowther CA. Prenatal administration of progesterone for preventing preterm birth in women considered to be at risk of preterm birth. Cochrane Database Syst Rev. 2013 Jul 31;2013(7):CD004947. doi: 10.1002/14651858.CD004947.pub3. PMID 23903965
- See also: Gestation-specific Infant Mortality: 2012 — https://www.ons.gov.uk/peoplepopulationandcommunity/healthandsocialcare/causesofdeath/bulletins/pregnancyandethnicfactorsinfluencingbirthsandinfantmortality/2014-10-15